CLINICAL TRIAL: NCT05335668
Title: Brain Circuitry Changes in Central Poststroke Pain: a Clinical and Neuroimaging Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-02640
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: CPP; Pain
MeSH Terms: conditions — Pain | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with central poststroke pain (Experimental): Patients with central poststroke pain
  Interventions: Procedure: Clinical Testing
- Patients without central poststroke pain (Experimental): Patients without central poststroke pain
  Interventions: Procedure: Clinical Testing
- healthy controls (Active Comparator): healthy volunteers
  Interventions: Procedure: Clinical Testing

INTERVENTIONS:
Procedure: Clinical Testing — Clinical testing for neurological deficits based on National Institute of Health Stroke Scale (NIHSS), objective sensory testing and pain assessment by quantitative sensory testing (QST) and quantitative pain drawings, 7T magnetic resonance imaging (MRI)

SUMMARY:
Central poststroke pain (CPP) is estimated to affect up to 10% of stroke patients and is one of the most difficult-to-treat conditions with a detrimental effect on patient's quality of life. So far, no drug has proven efficient to alleviate CPP and neuromodulation approaches including Deep Brain Stimulation (DBS) and motor-cortex stimulation have yielded mixed results with only a few patients experiencing long-term pain relief. To date, little is known about the pathophysiology of CPP. There is at present little evidence for a clear association between the specific location of lesions, clinical manifestation and phenomenology of pain as well as treatment response of CPP patients. Furthermore, the time delay between stroke occurrence and CPP occurrence is highly variable and the fact, that it is not immediate in the great majority of patients suggests that other factors contribute to the development of CPP. These factors have not been identified yet.

DETAILED DESCRIPTION:
Central poststroke pain (CPP) is estimated to affect up to 10% of stroke patients and is one of the most difficult-to-treat conditions with a detrimental effect on patient's quality of life. So far, no drug has proven efficient to alleviate CPP and neuromodulation approaches including DBS and motor-cortex stimulation have yielded mixed results with only a few patients experiencing long-term pain relief. To date, little is known about the pathophysiology of CPP. There is at present little evidence for a clear association between the specific location of lesions, clinical manifestation and phenomenology of pain as well as treatment response of CPP patients. Furthermore, the time delay between stroke occurrence and CPP occurrence is highly variable and the fact, that it is not immediate in the great majority of patients suggests that other factors contribute to the development of CPP. These factors have not been identified yet.

The objective of this research project is to correlate clinical aspects of CPP (pain phenomenology) with magnetic resonance image (MRI)-based findings, especially metabolic changes and functional reorganization processes captured by functional MRI and MR spectroscopy. A better understanding of the underlying pathophysiological mechanism of CPP and its involved neuronal networks are mandatory for any future therapeutic approach to treat this difficult condition. The discovery of a potential image-based biomarker could serve to help identify patients early who are at risk of developing CPP. Furthermore, the findings may help identify prognosticators of different forms of CPP treatments (e.g. biofeed-back, neuromodulation approaches, medication) in the future.

ELIGIBILITY:
Inclusion Criteria patients:

* Patients with a haemorrhagic or ischemic stroke affecting the somatosensory system as defined by both CT or MRI and clinical criteria
* Patient age between 18-75 years
* Signed written informed consent

Exclusion Criteria patients:

* Secondary stroke due to a cerebral vascular malformation or tumor
* Patients with aphasic syndromes and impaired verbal communication, complete sensory-motor hemi-neglect and restrictions of the ability to report on their pain and cooperate during sensory testing
* Patients with severe stroke NIHSS > 14 and or Modified Rankin Scale (MRS) > 3
* History of severe myelopathy or polyneuropathy with clinical sensory deficits and history of neuropathic pain
* Widespread stroke size due to internal carotid artery-occlusion or more than one main territory (anterior, middle or posterior cerebral artery)
* Contraindication for 7T MRI (metallic implant, tattoo, claustrophobia, etc.)
* In case of women < 45 years of age: pregnancy

Inclusion Criteria for healthy volunteers

* Informed consent as documented by signature
* Age: ≥18 years and ≤ 75 years

Exclusion criteria for healthy volunteers

* Pregnancy and breastfeeding
* Contraindication for 7T MRI (metallic implant, tattoo, claustrophobia, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between cerebral connectivity patterns | Day 30 after inclusion
  Correlation between cerebral connectivity patterns at rest during pain-processing tasks based on functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Pollo, MD, Principal Investigator — Inselspital Bern, Department of Neurosurgery
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowsher D. Central pain: clinical and physiological characteristics. J Neurol Neurosurg Psychiatry. 1996 Jul;61(1):62-9. doi: 10.1136/jnnp.61.1.62. PMID 8676164
- [Background] Bowsher D, Leijon G, Thuomas KA. Central poststroke pain: correlation of MRI with clinical pain characteristics and sensory abnormalities. Neurology. 1998 Nov;51(5):1352-8. doi: 10.1212/wnl.51.5.1352. PMID 9818859
- [Background] Karahanoglu FI, Van De Ville D. Transient brain activity disentangles fMRI resting-state dynamics in terms of spatially and temporally overlapping networks. Nat Commun. 2015 Jul 16;6:7751. doi: 10.1038/ncomms8751. PMID 26178017
- [Background] Preti MG, Bolton TA, Van De Ville D. The dynamic functional connectome: State-of-the-art and perspectives. Neuroimage. 2017 Oct 15;160:41-54. doi: 10.1016/j.neuroimage.2016.12.061. Epub 2016 Dec 26. PMID 28034766